CLINICAL TRIAL: NCT05789914
Title: Peking University School of Stomatology
Brief Title: The Efficacy of Guided Tissue Regeneration With Extracellular Matrix Scaffold of Small Intestinal Submucosa (SIS) Membrane: a Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKUSSIRB-202384005
Record Dates: First submitted 2023-03-01; First posted 2023-03-29 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Guided Tissue Regeneration; Extracellular Matrix Scaffold of Small Intestinal Submucosa
Keywords: guided tissue regeneration; Small Intestinal Submucosa; Randomized Controlled Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Small Intestinal Submucosa Membrane (Experimental)
  Interventions: Procedure: Flap surgery+bone graft+guided tissue regeneration
- Bio-guide (Active Comparator)
  Interventions: Procedure: Flap surgery+bone graft+guided tissue regeneration

INTERVENTIONS:
Procedure: Flap surgery+bone graft+guided tissue regeneration — after flap elevation and debridement, intrabony defect was filled with Bio-Oss and covered with membrane.

SUMMARY:
The most commonly used barrier membrane material in guided tissue regeneration is absorbable collagen membrane. Although the collagen membrane has a good barrier effect, it lacks the growth factors needed for periodontal tissue regeneration, which affects the effect of collagen membrane on periodontal tissue regeneration. Extracellular Matrix Scaffold of Small Intestinal Submucosa (SIS) Membrane is a novel absorbable membrane that retains the extracellular matrix structure and is conducive to vascular ingrowth and tissue repair. The in vitro study showed that SIS membrane had excellent biocompatibility and certain antibacterial effect. Preclinical study also showed that SIS membrane significantly promoted the differentiation of bone marrow mesenchymal stem cells into osteoblasts, and promoted bone regeneration more effectively than collagen mechanism materials. SIS membrane can be used in soft tissue wound repair, guided bone regeneration, site preservation and other surgeries, and has achieved good therapeutic effects. However, whether the application of SIS membrane can achieve good therapeutic effect on periodontal guide tissue regeneration is still unclear. Therefore, in this study, the effects of guide tissue regeneration with collagen membrane and SIS membrane were compared through a randomized controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis patients with stage III to IV, grade C had one or more intrabony defects with a depth of ≥3 mm; PD≥5mm after initial periodontal therapy.

Exclusion Criteria:

* smokers, pregnant female, other systematic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical attachment loss | Baseline and 6 months after surgery
  before and 6 months after surgery, examine the changes of CAL
clinical attachment loss | baseline and 12 months after surgery.
  before and 12 months after surgery, examine the changes of CAL

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Hospital of stomatology, Beijing, Beijing Municipality, China